CLINICAL TRIAL: NCT00186680
Title: Selection of CD34+THY-1 Positive Cells From Peripheral Blood Cells Procured for Autologous Hematopoietic Support Following High Dose Treatment With BCNU, Cyclophosphamide & Cisplatin for Stage IV Breast Cancer & Limited Prior Treatment
Brief Title: CD34 Selection of the Peripheral Blood Stem Cell Graft for Autologous Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Ginna Laport, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT86; BMT86; NCT00186680
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: high dose chemo then auto hematopoietic cell transplant

SUMMARY:
Evaluate the feasibility and safety of autologous transplantation of CD34+Thy-1+ hematopoietic stem cells afer high dose marrow ablative chemotherapy in patients with breast cancer.

DETAILED DESCRIPTION:
Selection of CD34+THY-1 Positive Cells From Peripheral Blood Cells Procured for Autologous Hematopoietic Support Following High Dose Treatment with BCNU, Cyclophosphamide & Cisplatin for Stage IV Breast Cancer & Limited Prior Treatment

ELIGIBILITY:
Inclusion Criteria:- stage IV breast cancer

* primary breast cancer does not express CD34+
* adequate organ function
* no evidence of active infection Exclusion Criteria:- chemotherapy within 4 weeks
* CNS disease

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 1996-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety

SECONDARY OUTCOMES:
efficiency of mobilization
tumor contamination

CONTACTS AND LOCATIONS:
Overall Officials: Ginna Laport, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States